CLINICAL TRIAL: NCT07266103
Title: Building on Previous Evidence: A Mechanistic Clinical Trial of Personalized rTMS for Chronic Pain
Brief Title: Mechanistic Study of Personalized rTMS in Chronic Pain
Acronym: PRECISE-Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Principal investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20230076-4
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
Keywords: pain; TMS-EEG; rTMS
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: When 50% of inclusion is completed, a preplanned interim futility analysis is scheduled to examine safety and the main outcome.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator : Classical rTMS (Active Comparator): The patients will receive repetitive transcranial magnetic stimulation according to the classical treatment
  Interventions: Device: Classical repetitive trancranial magnetic stimulation to M1
- Experimental: Personalized Target Arm (Experimental): The patients will receive repetitive transcranial magnetic stimulation (rTMS) to target showing the optimal connectivity during the TMS-EEG assessment one week before starting the treatment
  Interventions: Device: Personalized Target Arm

INTERVENTIONS:
Device: Classical repetitive trancranial magnetic stimulation to M1 — The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds with an interval of twenty seconds between trains will be delivered, as traditionally performed. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes.
  Arms: Active Comparator : Classical rTMS
Device: Personalized Target Arm — The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds will be delivered with an interval of twenty seconds between trains. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes. The rTMS will be delivered to the optimal target
  Arms: Experimental: Personalized Target Arm

SUMMARY:
Previous research has demonstrated that repetitive magnetic brain stimulation can be an effective adjunctive treatment for several conditions, including chronic pain. However, current stimulation protocols are typically standardized and do not account for individual variability in brain function. This uniform, one-size-fits-all approach results in only about 40% of patients experiencing meaningful clinical benefit, while the remainder show little to no improvement. To address this limitation, the present study will investigate how magnetic stimulation can be tailored to individuals with chronic pain. By analyzing each participant's brain signals prior to treatment, we aim to personalize stimulation parameters to better match individual neural characteristics and potentially enhance therapeutic outcomes. The design of this study builds directly on the findings of a previous clinical trial.

DETAILED DESCRIPTION:
This study builds directly on previous clinical findings identifying four cortical targets-primary motor cortex (M1), anterior cingulate cortex (ACC), dorsolateral prefrontal cortex (DLPFC) and the posterior insula (PSI)-as exhibiting neurophysiological properties potentially useful for guiding individualized repetitive transcranial magnetic stimulation (rTMS) target selection. Earlier results demonstrated that chronic pain patients with low alpha-band intertrial coherence (ITC) over M1 were more likely to respond to stimulation of M1, whereas patients with high alpha-band ITC showed a greater likelihood of responding to stimulation of PSI, ACC or DLPFC. These findings suggest that specific electroencephalography (EEG) connectivity markers may help predict the cortical target most likely to provide therapeutic benefit for an individual patient.

Building on this evidence, the present trial will classify participants according to their pre-treatment transcranial magnetic stimulation-electroencephalography (TMS-EEG) connectivity profiles and assign treatment to the cortical region with the highest predicted probability of clinical response.

A total of 90 patients with chronic pain will be enrolled in a double-blind, randomized, two-parallel-arm clinical trial comparing the analgesic effects of individualized target selection with those of the standard rTMS protocol. Participants will be randomized 1:1 to:

* Individualized targeting, in which the rTMS site is selected based on each participant's TMS-EEG connectivity profile
* Standard stimulation, representing the conventional rTMS approach for pain relief.

At baseline, participants will complete standardized questionnaires and undergo neurophysiological assessments, including single-pulse TMS-EEG for target classification. The induction phase will then begin, consisting of five consecutive daily rTMS sessions delivered Monday through Friday. Each session lasts 30 minutes, including 15 minutes of active stimulation.

The induction phase will be followed by a 7-week maintenance phase, during which participants receive one rTMS session per week (seven sessions in total). At the end of the maintenance phase, all outcome measures will be reassessed to evaluate treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic pain (present most of the days for more than 3 months).
* Pain with a mean pain intensity between 3-9 on a 0-10 pain scale (where 0 means no pain and 10 means the worst pain imaginable).
* Speak and understand English or Danish

Exclusion Criteria:

* Pregnant or breastfeeding
* Current uncontrolled major depression as the main diagnosis
* Current history of substance abuse
* Lack of ability to cooperate, to fully understand the protocol or any difficulty in filling out questionnaires (e.g., due to language or cognitive problems)
* Formal contraindications to TMS application (presence of epilepsy, cranial implanted ferromagnetic devices, e.g., intracranial neurostimulator or cochlear implants, tattoos with metal ink on the face or permanent make up with metal in the face )
* Unable to answer the "Transcranial Magnetic Stimulation Adult Safety Screen" screening questionnaire.
* Participation in other research protocols within 1 month before the inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual analogue scale) | Visual analogue scale will be assessed before treatment, after 2 months, and again after 3 months. Responders are those with ≥30% pain reduction at the end of maintenance compared to average pain intensity the week before baseline assessment.
  The '0' represents 'no pain' at all, and '100' represents the 'worst possible pain' that the individual can imagine.

SECONDARY OUTCOMES:
Quality of life (EQ-5D) | Quality of life changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  Quality of life (EQ-5D) is a standardized measure of health-related quality of life. This is the value derived from the 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ-5D-5L is a scale from 0 to 100, where 100 is the best health imaginable.
Patients' Global Impression of Change | Patients' Global Impression of Change will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment
  The questionnaire assesses the individual's impression of change after an intervention. Minimum value: 1 = "Very much worse" and Maximum value: 7 = "Very much improved"
Short Brief Pain Inventory | Short Brief Pain Inventory changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning
Connectivity analysis | Connectivity changes will be investigated before the treatment and immediately after 2 months of treatment.
  Electroencephalography recorded during single pulses of transcranial magnetic stimulation will be used to evaluate brain connectivity. Global mean field power, local mean field power, inter-trial coherence and event-related strectral perturbation will be the main outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico De Martino, Principal Investigator — Aalborg University

IPD SHARING:
Plan to Share IPD: No